CLINICAL TRIAL: NCT00687700
Title: A Study to Investigate the Relative Pharmacological Activity of Aninhaled B2-agonist/Anticholinergic Dual Pharmacophore Inhealthy Volunteers
Brief Title: A Study to Investigate the Pharmacology of a Dual Pharmacophore in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Theravance Biopharma (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Purpose: Treatment
Other Study IDs: MAB110553
Record Dates: First submitted 2008-05-28; First posted 2008-06-02 (Estimated); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: propranolol; B2-agonist,; B-antagonist,
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — batefenterol; Propranolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All subjects (Experimental): Eligible subjects will receive GSK961081 (400 micrograms or 1200 micrograms), GSK961081 matching placebo, propranolol (80 milligrams) and propranolol matching placebo in five treatment sessions through ten different crossover treatment sequences. There will be a washout period between treatment sessions of 7 to 14 days.
  Interventions: Drug: GSK961081; Drug: GSK961081 matching placebo; Drug: Propranolol; Drug: Propranolol matching placebo

INTERVENTIONS:
Drug: GSK961081 — GSK961081 multidose dry powder inhaler (Diskus inhaler) will be available with dosing strengths of 400 micrograms and 1200 micrograms administered once daily in the morning.
Drug: GSK961081 matching placebo — GSK961081 matching placebo multidose dry powder inhaler (Diskus inhaler) will be available to be administered once daily in the morning.
Drug: Propranolol — Propranolol over encapsulated tablet will be available with dosing strengths of 40 milligrams administered orally with 240 milliliters of water.
Drug: Propranolol matching placebo — Propranolol matching placebo over encapsulated tablet will be available to be administered orally with 240 milliliters of water.

SUMMARY:
Study will investigate the pharmacodynamics of a dual pharmacophore in which a combination of GSK961081 and Propanolol is used to give a total effect of bronchodilation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males aged between 18 and 50 years.
* Body mass index within the range 19-29.9 kg/m2.
* FEV1 ≥ 80% predicted and a FEV1/ Forced Vital Capacity (FVC) ratio ≥ 0.7
* Signed and dated written informed consent is obtained from the subject
* The subject is able to understand and comply with the protocol requirements, instructions and protocol-stated restrictions.
* The subject has an increase in sGAW of ≥15% over pre-dose baseline within 2 h of administration of 400 µg salbutamol by MDI inhaler at screening or in the 3 months before screening.
* The subject has an increase in sGAW of ≥25% over pre-dose baseline within 2 h following 80 µg ipratropium bromide at screening or in the 3 months before screening.
* Subjects who are current non-smokers who have not used any tobacco products in the 6-month period preceding the screening visit and have a pack history of ≥ 10 pack years.

Exclusion Criteria:

* Any clinically relevant abnormality identified at the screening medical assessment (physical examination/medical history), clinical laboratory tests, or ECG (12-lead or Holter).
* A history of respiratory disease (i.e. history of asthmatic symptoms).
* Clinically significant abnormal 12 lead ECG at
* A subject in whom ipratropium bromide, salbutamol or propranolol are contraindicated.
* A supine blood pressure that is persistently higher than 140/90 millimetres of mercury (mmHg) at screening.
* A supine mean heart rate outside the range 45-90 beats per minute (bpm) at screening.
* The subject has donated a unit of blood within the 56 days or intends to donate within 56 days after completing the study.
* The subject is currently taking regular (or course of) medication whether prescribed or not (with the exception of contraceptives, including vitamins and herbal remedies such as St John's Wort.
* The subject has used prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (which ever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and medical monitor the medication will not interfere with the study procedures or compromise subject safety.
* The subject has participated in a clinical study with a New Chemical Entity (NCE) within the past 3 months.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* The subject is infected with the Hepatitis B, Hepatitis C, or HIV virus.
* The subject has a positive pre-study urine cotinine/ breath carbon monoxide test, urine drug/urine alcohol screen.
* A history of regular alcohol consumption exceeding weekly intake of alcohol greater than 28 units for males, or an average daily intake of greater than 4 units.
* Are unable to use the inhaler correctly.
* The subject has a history of drug or other allergy, which, in the opinion of the Investigator, contraindicates their participation.
* The subject has had a lower respiratory tract infection within 4 weeks of study start.
* Subject is unable to perform the sGAW measurements

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2008-03-10 (Actual); Primary Completion 2008-05-27 (Actual); Study Completion 2008-05-27 (Actual)

PRIMARY OUTCOMES:
To assess the bronchodilation of single doses of GSK961081 over 24 hours following ß blockade with the ß antagonist propranolol as measured by sGaw in healthy subjects. | Up to 32 hours

SECONDARY OUTCOMES:
Assess safety of GSK961081 after single doses of it with&without ß blockade with propranolol as measured by specific indicators | Up to 71 days
Adverse events, clinical laboratory safety tests, FEV1, vital signs, 12-lead ECG parameters, blood glucose and serum potassium. | Up to 71 days
Propranolol and GSK961081blood levels to derive pharmacokinetics | Up to 32 hours
Assess systemic pharmacokinetics of GSK961081 and propranolol after single doses of both | Up to 32 hours

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Harrow, Middlesex, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study MAB110553 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/MAB110553?search=study&study_ids=MAB110553#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: MAB110553 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: MAB110553 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: MAB110553 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: MAB110553 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: MAB110553 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: MAB110553 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: MAB110553 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register